CLINICAL TRIAL: NCT01349296
Title: BARIS - BIBF1120 and RAD001 in Solid Tumors. A Phase I Trial to Evaluate the Safety and Tolerability of Combined BIBF 1120 and RAD001 in Solid Tumors and to Determine the Maximum Tolerated Dose (MTD) of the Combination
Brief Title: BIBF 1120 and RAD001 in Solid Tumors - Phase I
Acronym: BARIS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Cologne (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Principal Investigator, Prof. Dr. Juergen Wolf, Prof. Dr., Lung Cancer Group Cologne
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BARIS
Record Dates: First submitted 2011-05-05; First posted 2011-05-06 (Estimated); Last update posted 2016-05-20 (Estimated); Status verified 2016-05

CONDITIONS: Solid Tumors
Keywords: Solid Tumors
MeSH Terms: interventions — Everolimus; nintedanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BIBF 1120 + RAD001 (Experimental)
  Interventions: Drug: Everolimus + BIBF 1120

INTERVENTIONS:
Drug: Everolimus + BIBF 1120 — Dose level 1: 1x 5mg Everolimus/d + 2x 150mg BIBF 1120/d. Dose level 2: 1x 5mg Everolimus/d + 2x 200mg BIBF 1120/d. Dose level 3: 1x 10mg Everolimus/d + 2x 200mg BIBF 1120/d
  Other Names: Everolimus, RAD001, Afinitor, BIBF 1120

SUMMARY:
BIBF1120 and RAD001 in solid tumors

DETAILED DESCRIPTION:
A phase I trial to evaluate the safety and tolerability of combined BIBF 1120 and RAD001 in solid tumors and to determine the maximum tolerated dose (MTD) of the combination

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically proven solid tumor disease after failure of standard therapy regimen(s)
2. Age > 18 years.
3. ECOG performance status 0 to 1.
4. Life expectancy of at least 12 weeks.
5. Subjects with at least one measurable (CT or MRI) lesion.
6. Adequate bone marrow, liver and renal function as assessed by the following laboratory requirements conducted within 7 days prior to screening:

   * Hemoglobin > 9.0 g/dl
   * Absolute neutrophil count (ANC) >1,500/mm3
   * Platelet count ³ 100,000/μl
   * Total bilirubin within normal limits
   * ALT and AST < 1.5 x upper limit of normal ( or < 2.5 x upper limit of normal in patients with liver involvement)
   * PT-INR/PTT < 1.5 x upper limit of normal [Patients who are being therapeutically anticoagulated with an agent such as coumadin or heparin will be allowed to participate provided that no prior evidence of underlying abnormality in these parameters exists.]
   * Serum creatinine < 1.5 x upper limit of normal or creatinine clearance (CrCl) ≥ 50 ml/min calculated by either Cockcroft-Gault or by 24 hours urine collection
7. More than 14 days since previous chemotherapy, radiotherapy and surgery
8. Negative urine or serum HCG in women of childbearing potential
9. Signed and dated informed consent before the start of specific protocol procedures

Exclusion Criteria:

1. Limited number of prior lines of treatment (including surgery and radiotherapy, if part of the standard therapy of the respective tumor entity)
2. Prior treatment with BIBF 1120 or any other VEGFR inhibitor (bevacizumab is allowed)
3. Prior treatment with RAD001 or any other mTOR inhibitor
4. Known hypersensitivity to the trial drugs, to their excipients or to contrast media
5. Chemo-, hormono-, radio-(except for brain and extremities) or immunotherapy or therapy with monoclonal antibodies or small tyrosine kinase inhibitors within the past 2 weeks prior to treatment with the trial drugs
6. Persistence of clinically relevant therapy related toxicity from previous chemo and/or radiotherapy
7. Active brain metastases (e.g. stable for <4 weeks, no adequate previous treatment with radiotherapy, symptomatic, requiring treatment with anticonvulsants; dexamethasone therapy will be allowed if administered as stable dose for at least one month before trial drug administration) or leptomeningeal metastases (documented by lumbar puncture)
8. History of cardiac disease: congestive heart failure >NYHA class 2; active coronary artery disease (CAD), (MI more than 6 mo prior to study entry is allowed); cardiac arrhythmias requiring antiarrhythmic therapy (beta blockers or digoxin are permitted) or uncontrolled hypertension
9. Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of BIBF1120 or RAD001 (e.g. ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome or small bowel resection)
10. History of HIV infection or previously seropositive for the virus
11. History of Hepatitis B or/and C or previously seropositive for the Hepatitis B or/and C virus
12. Radiographic evidence of cavitary or necrotic tumors
13. Centrally located tumors with radiographic evidence (CT or MRI) of local invasion of major blood vessels
14. Treatment with other investigational drugs or treatment in another clinical trial within the past 30 days before start of therapy or concomitantly with the trial
15. Patients with seizure disorder requiring enzyme-inducing antiepileptics
16. Therapeutic anticoagulation (except low-dose heparin and/or heparin flush as needed for maintenance of an indwelling intravenous devise) or antiplatelet therapy (except for low-dose therapy with acetylsalicylic acid ≤325mg per day)
17. Major injuries within the past 10 days prior to start of study treatment with incomplete wound healing and/or planned surgery during the on-treatment study period
18. Evidence or history of bleeding diasthesis or thrombosis, and known inherited predisposition to bleeding or thrombosis
19. Proteinuria CTC AE grade 2 or greater
20. Active serious infections
21. Patients undergoing renal dialysis
22. Previous or concurrent cancer that is distinct in primary site or histology from the cancer being evaluated in this study EXCEPT cervical carcinoma in situ, treated basal cell carcinoma, superficial bladder tumors [Ta, Tis & T1] or any cancer curatively treated > 3 years prior to study entry
23. Serious illness or concomitant non-oncological disease such as neurologic, psychiatric, infectious disease or active ulcers (gastrointestinal tract, skin) or laboratory abnormality that may increase the risk associated with study participation or study drug administration and in the judgment of the investigator would make the patient inappropriate for entry into the study
24. Patients who are sexually active and unwilling to use a medically acceptable method of contraception (e.g. such as implants, injectables, combined oral contraceptives, some intrauterine devices or vasectomized partner for participating females, condoms for participating males) during the trial and for at least three months after end of active therapy
25. Pregnancy or breast feeding
26. Psychological, familial, sociological or geographical factors potentially hampering compliance with the study protocol and follow-up schedule
27. Active alcohol or drug abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2012-07; Primary Completion 2014-10 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose (MTD) of RAD001 in combination with BIBF 1120 (150mg bid or 200mg bid) (endpoint: dose-limiting toxicities) | Every visit
  Documentation an estimation of adverse events
To evaluate the tolerability of BIBF1120 and RAD001 in combination (endpoints: assessment of adverse events (AEs) according to CTC-AE V4.0) | Every visit during the study
  Documentation an estimation of adverse events

SECONDARY OUTCOMES:
To evaluate the clinical efficacy of the combination descriptively (endpoints: RR, progression free survival (PFS), overall survival (OS)) | Baseline and every six weeks during the study, after study every 6 months
  CT will be done for evaluation of RR and PFS on day 57 and then every 6 weeks until progression.
  For overall survival a telephone call every six months after study is continuation will be done
To analyze individual BIBF1120 pharmacokinetic (PK) parameters at steady-state (ss) of monotherapy and PK parameters of both BIBF1120 and RAD001 at ss of combination | day 14, day 29
  Blood collection for pharmacokinetic analysis
To assess changes in tumor vasculature a) early under BIBF1120 monotherapy, b) at ss of BIBF1120 monotherapy and c) at ss of combination therapy using dynamic contrast-enhanced MRI (DCE-MRI) (endpoints: IAUC, Ktrans, Kep, Ve) | baseline, day 3, day 14, day 29
  DCE MRI will be done
To correlate the clinical outcome with FGFR1-amplification status (endpoints: see above for clinical parameters) | Screening
  Documentation of histology

CONTACTS AND LOCATIONS:
Overall Officials: Juergen Wolf, Prof., Principal Investigator — University Hospital of Cologne
Locations (1):
- University Hospital of Cologne, Cologne, North Rhine-Westphalia, Germany